CLINICAL TRIAL: NCT05654311
Title: The Relationship Between Emergence Agitation and Electroencephalogram in Young Adults Undergoing Nasal Surgery Under General Anesthesia
Brief Title: Performance of EEG During Emergence Agitation in Nasal Surgery.
Status: Recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate Professor, Gangnam Severance Hospital
Other Study IDs: 3-2022-0351
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Nasal Surgery
Keywords: general anesthesia; electroencephalogram; emergence agitation; sevoflurane
MeSH Terms: conditions — Emergence Delirium | interventions — Nasal Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nasal surgery — Nasal surgery under general anesthesia using inhalational agent (sevoflurane)

SUMMARY:
The purpose of the study is to evaluate the relationship between perioperative electroencephalogram and emergence agitation in the nasal surgery. Previous studies showed that low frequency band wave activity increased during emergence delirium in pediatric patients. It is still not enough to explain the relationship between emergence agitation and electroencephalogram in adults. Researchers will demonstrate the relationship between parameters related electroencephalogram and emergence agitation in adults undergoing nasal surgery.

DETAILED DESCRIPTION:
Researchers use Sedline to perform perioperative EEG measurements of young adult patients undergoing nasal surgery under general anesthesia with sevoflurane. Emergence agitation occurrence and EEG patterns are observed.

The researchers record the patient's sex, type of surgery, pre-education on emergence agitation, preoperative hospital anxiety and depression scale (HADS), postoperative pain, amount of analgesics administered in the surgery/recovery room, and PACU time. Investigators check the correlation between EEG and perioperative variables. Investigators also compare EEG and perioperative variables for those who were given an explanation of emergence agitation and those who were not.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19-55 years who are undergoing nasal surgery under general anesthesia using inhalational agent

Exclusion Criteria:

* CNS disease (ex.dementia, stroke, brain tumor, psychological disorder..)
* unable to communicate
* general anesthesia history within 6 months
* disagree to participate in study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study collects subjects from a tertiary university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-10-26 (Estimated); Study Completion 2024-10-26 (Estimated)

PRIMARY OUTCOMES:
EEG band relative power measured in the frontal lobe | From the cessation of sevoflurane inhalation to the extubation of tracheal tubes
  relative power of each brain waves : Original frontal EEG waves using 4 channel sedline (Masimo, Irvine, CA, USA) sensor will processed by FFT(fast Fourier transform). Each band is as follows.: Delta: 1-4 Hz Theta: 4-8 Hz Alpha: 8-13 Hz Beta: 13-30 Hz.
occurrence of emergence agitation | From the cessation of sevoflurane inhalation to transfer to the recovery room
  Emergence agitation occurrence : RASS(Richmond Agitation Sedation Score) is 10 scaled (-5~+4) score to assess sedation/agitation level; 0 is a calm state, and a value less than 0 means a sedation state.

SECONDARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) | 1 day before surgery (after admission)
  A self-assessment scale, brief, clinically useful measure of anxiety and depression symptoms. It can be used to diagnose depression in people with significant physical ill-health.
VAS (Visual Analogue Scale) | during 30 minutes after PACU admission
  Using a ruler, it is 11 scaled (0-10) score to assess pain.
Effect of preoperative education on emergence agitation | up to 6 months after completion of the study
  Investigate the relationship between preoperative emergence agitation explanation and occurrence of emergence agitation

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital Yonsei University College of Medicine, Seoul, South Korea